CLINICAL TRIAL: NCT07326956
Title: Efficacy of Core Stability Training on Endurance, Kinetic Chain Function, and Dynamic Balance in Healthy Adult Soccer Players: A Randomized Controlled Trial
Brief Title: Efficacy of Core Stability Training on Endurance, Kinetic Chain Function, and Dynamic Balance in Soccer Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Shibili Nuhmani, Assistant professor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-PGS-2025-03-0529
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: The Study Investigates the Efficacy of Core Stability Training on Core Endurance and Kinetic Chain Function and Dynamic Balance in Healthy Adult Soccer Players
Keywords: Keywords: core stability, endurance, kinetic chain, athletes, soccer.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core training group (Experimental): This group will receive core stability training + their regular soccer training
  Interventions: Other: Core stability exercises; Other: Regular soccer training
- control group (Active Comparator): this group will continue their usual soccer training
  Interventions: Other: Regular soccer training

INTERVENTIONS:
Other: Core stability exercises — exercises for the trunk, pelvic, and hip muscles
  Arms: core training group
Other: Regular soccer training — the routine exercises performed regularly by soccer players

SUMMARY:
Background: The core has two functions, both critical to soccer performance. The first is to provide proximal stability, allowing efficient mobility at the distal parts. This function requires a submaximal contraction of core muscles for as long as the movement takes. It was reported that core endurance is the construct most closely representing this function. The second function is generating and transferring forces from one extremity to another. This function operates via the kinetic chain theory, which implies that various body parts are connected through myofascial kinetic chains, and that a defect in one part of the chain can lead to faulty mechanics and balance, potentially causing injuries in other parts of that chain.

Aim: To investigate the efficacy of core stability training on core endurance, lower limb kinetic chain function, and lower limb dynamic balance in professional, healthy young adult soccer players.

Methods: This is a randomized, controlled trial with a parallel, two-arm, pre- and post-design. After screening for eligibility and obtaining participants' consents, at least 28 male and female soccer players will be randomly assigned to intervention and control groups and tested before and after eight weeks of core training intervention. The outcome measures include the Sport-specific Endurance Plank test, the Closed Kinetic Chain Lower Extremity Stability test, and the modified Star Excursion Balance test.

Data Analysis: The Shapiro-Wilk test, Q-Q plots, and Box plots will be used to evaluate the normality of the data. Lavan's test will check the homogeneity of variances. Based on the normality results, parametric or non-parametric tests will be implemented to compare within and between groups. A P-value of <0.05 will be used to reflect the significance of the results. An intention-to-treat (ITT) analysis will be employed to address potential missing data.

Keywords: core stability, endurance, kinetic chain, athletes, soccer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, young adult soccer players of both genders between 18 and 35 years.
* Normal Body mass index (BMI) according to the World Health Organization (WHO) guidelines (18.5-24.9).
* Normal waist circumference (<88 cm for women and < 102 cm for men).

Exclusion Criteria:

* As reported by participants, they will be excluded if they have a history of:

  * Chronic diseases (e.g., cardiovascular diseases, diabetes mellitus, hypertension).
  * Peripheral vascular diseases (e.g., deep venous thrombosis).
  * Systemic diseases (e.g., rheumatoid arthritis, lupus erythematosus)
  * Limbs or trunk trauma, injuries, fractures, or surgeries that required medical attention in the past six months.
  * Concussion.
  * Neurological deficits or symptoms (e.g., numbness, referred to pain to the lower limbs, burning sensation).
  * The use of any medications that might affect the testing procedure and training.
  * Physical pain (e.g., back pain, limb pain).
  * Red flags (e.g., sudden loss of weight, night sweats, or fever).
  * Pregnancy and post-partum (1 year)
* Upon inspection and palpation by the primary researcher, participants will be excluded if they have:

  * Biomechanical abnormalities or deformities in the upper or lower limbs.
  * Swelling/ edema
  * Leg length discrepancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Sport-specific Endurance Plank test | 60 seconds
  Participants will start with a standard prone plank position on a bench supported on their elbows and feet. They must keep their head, torso, pelvis, and heels in a straight line and their elbows aligned vertically with their shoulders. While maintaining this position for 60 seconds (s), they will perform several tasks consecutively: (1) raise their right arm for 15 s, then lower it and raise their left arm for 15 seconds, then lower it down; (2) lift the right leg (in a straight position) for 15 s, then lower it and lift the left leg for 15 seconds and lower it down; (3) raise the right arm and left leg (diagonally) for 15 s and lower them down; (4) raise the left arm and right leg (diagonally) for 15 s and lower them down; (5) keep the prone plank position for 30s. Then, participants will repeat the same steps (1-5) until the prone plank position cannot be maintained.
Closed Kinetic Chain Lower Extremity Stability Test | 15 seconds
  First, participants will be asked to lie on the floor mat in a prone plank position; their feet will be apart at shoulder width. While maintaining the prone plank position with their body kept in a straight line, participants will be asked to start crossing their legs alternately as fast as possible for 15 seconds. The Assessor will start the stopwatch, pre-setted for 15 seconds when the participants start moving. The assessor will simultaneously and manually count the number of successful crosses each participant can make during those 15 seconds. A successful cross is defined as participants touching, with their moving foot, the floor at the lateral side of their stationary foot and then fully returning to the starting position.

SECONDARY OUTCOMES:
The Modified Star Balance Excursion Test | 10 minutes
  The floor will be taped with three crossing lines. Participants will be asked to stay barefoot and to stand upright with one foot (foot of the testing limb) positioned in the middle of the grid. The most distal part of the big toe of the stance leg should be placed just at the crossroad between the three lines. The position of the stationary foot should remain constant throughout the whole testing procedure. Moreover, participants' hands shall remain on their hips throughout the test to focus on the lower limb performance. Participants will then be asked to reach as far as possible with the other limb in each of the three directions. They should touch (without weight bearing) the line where they can maximally reach by the most distal part of the big toe and return to the starting position without losing their balance. Using a tape measure, the assessor will measure and record the distance (in centimeters) reached.

IPD SHARING:
Plan to Share IPD: No
To ensure the confidentiality of our participants' information.